CLINICAL TRIAL: NCT04110093
Title: The Efficacy and Safety of Regorafenib Plus PD-1 Inhibitor as Third-line Therapy in Advanced Colorectal Cancer Patients
Brief Title: Regorafenib Plus PD-1 Inhibitor in Patients With Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Yuan-Sheng Zang, Head of Medical Oncology Department, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZ-REGONIVO
Record Dates: First submitted 2019-09-28; First posted 2019-10-01 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Cancer; Immunotherapy
Keywords: Colorectal Cancer; Immunotherapy; Regorafenib; Nivoluamb; microsatellite stable
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy Combination treatment (Experimental): All colorectal cancer patients received regorafenib plus PD-1 inhibitor
  Interventions: Drug: Regorafenib and PD-1 inhibitor

INTERVENTIONS:
Drug: Regorafenib and PD-1 inhibitor — All Colorectal cancer patients received regorafenib (80mg qd d1-d21,q4w) and PD-1 inhibitor. The patients could receive one type of PD-1 inhibitors according to oneself circumstance consideration including nivolumab (3mg/kg, ivgtt, q2w), Carelizumab (200mg, ivgtt, q3w), Sintilimab (200mg, ivgtt, q3w), Toripalimab(240mg ivgtt, q3w).

SUMMARY:
This study is intended to evaluate efficacy and safety of the combination of regorafenib and nivolumab as third-line or later therapy in patients with microsatellite stable (MSS) colorectal cancer (CRC).

ELIGIBILITY:
Inclusion Criteria:

* Advanced Colorectal Cancer diagnosed histologically;
* Patients with microsatellite stable (MSS)
* Patients have no any standard choice after multiple line of therapy( ≥ 2 lines);
* Expected survival ≥ 3 month;
* ECOG / PS score: 0-2, and the main organ function to meet the following criteria: HB ≥ 90g / L, ANC ≥ 1.5 × 109 / L, PLT ≥ 80 × 109 / L,BIL <1.5 times the upper limit of normal (ULN); Liver ALT and AST <2.5 × ULN and if liver metastases, ALT and AST <5 × ULN; Serum Cr ≤ 1 × ULN, endogenous creatinine clearance ≥50ml/min

Exclusion Criteria:

* Patient still has standard treatment therapy based on NCCN guidance;
* Patient can not comply with research program requirements or follow-up;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 2 months
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission.
Progress Free Survival | Evaluation of tumor burden based on RECIST criteria until first documented progress through study completion, an average of 2 months
  Time from treatment beginning until disease progression

SECONDARY OUTCOMES:
Overall Survival | From date of treatment beginning until the date of death from any cause, through study completion, an average of 1 months
  Time from treatment beginning until death from any cause
Adverse Effect | Through study completion, an average of 1 months
  Incidence of Treatment-related adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Shanghai Changzheng Hospital, Shanghai, China